CLINICAL TRIAL: NCT05439980
Title: Development of Effective Resources for Phosphate Education for Children and Families With Chronic Kidney Disease: Hearing the Patient Voice
Brief Title: Improving Phosphate Control in Children With CKD
Acronym: IMPACT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Rukshana Shroff1, Professor, Great Ormond Street Hospital for Children NHS Foundation Trust
Other Study IDs: 21BO24
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Chronic Kidney Diseases; Hyperphosphatemia; Pediatric Kidney Disease; CKD-MBD; Chronic Kidney Disease-Mineral and Bone Disorder
Keywords: Dietary phosphate; Phosphate knowledge questionnaire
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CKD aged 8-<13 years: 8-<13 years n = 25
  Interventions: Other: Knowledge questionnaire; Other: Focus groups
- CKD aged 13-18 years: 13-18 years n = 25
  Interventions: Other: Knowledge questionnaire; Other: Focus groups
- Parents/caregivers: Parent/caregivers of children and young people with CKD 4-5D n=50
  Interventions: Other: Knowledge questionnaire; Other: Focus groups

INTERVENTIONS:
Other: Knowledge questionnaire — Completion of a questionnaire at baseline
Other: Focus groups — structured interviews

SUMMARY:
Research goals:

To explore the views and baseline knowledge of children and young people (CYP) with CKD and their caregivers to develop effective phosphate educational materials (PEM), adapted for age, and acknowledging different learning styles

DETAILED DESCRIPTION:
Background and Rationale

Background:

CKD mineral and bone disorder (CKD-MBD) can lead to debilitating skeletal complications, fractures, poor growth and vascular calcification, and remains one of the most challenging areas of CKD management. Serum phosphate and related measures of MBD, including Fibroblast Growth Factor 23 (FGF23) and parathyroid hormone (PTH), are raised in CKD and causally associated with adverse outcomes including vascular damage and calcification, left ventricular hypertrophy and renal bone disease. Reduction in dietary phosphate intake and regular intake of phosphate binder medications is required for optimal phosphate control but is extremely challenging, leading to poor adherence in a significant number of patients. The International Paediatric Dialysis Network Registry reports that in over 900 children on PD, 45% had high serum phosphate levels, with the prevalence of hyperphosphataemia increasing to 80% in adolescents.

Paediatric renal dietitians are responsible for educating families about dietary phosphate intake: limiting foods high in organic phosphate as well as avoiding the "hidden" inorganic phosphate from food additives, without compromising nutritional adequacy. Phosphate educational material (PEM) have been developed primarily for adults but dietary adherence is less than 50%, and is similarly low in children. Not only must children understand how to reduce their dietary phosphate intake but also how to use phosphate binder medication to reduce phosphate absorption from their foods and drinks. Adherence to binder medication is typically low due to poor palatability and the complexity of administration. Phosphate binder adherence is compounded by issues of access at school and psychological impacts, particularly during adolescence.

Educational interventions have mainly focused on the adult haemodialysis population with short-term follow-up. There are eight randomised controlled trials (RCTs) of using an educational intervention in adults with CKD or on dialysis which conclude that such interventions increased adherence compared to no intervention or routine standard care. A meta-analysis of adult RCTs also reported that educational initiatives can improve serum phosphate levels. Adult data has limited applicability to the management of hyperphosphataemia in CYP, as understanding and compliance with dietary restrictions will often be a joint responsibility between the CYP and their caregivers. There are very few studies assessing the success of educational programmes in paediatrics but, despite some showing an improvement in knowledge scores, interventions seem not to be associated with changes in serum phosphate or PTH. However, these studies had small sample sizes, were of short duration and learning patterns or factors influencing behaviour were not explored. Education strategies to balance dietary phosphate load to binder dose have been developed for children but require a high degree of patient motivation and do not account for the variable presence and bioavailability of inorganic and organic phosphate. The very high prevalence of hyperphosphataemia and its complications makes it clear that current management strategies are not effective and that alternative approaches are required to ensure optimal phosphate control.

Gaining feedback from children and their families about the challenges they face with phosphate control, as well as how they respond to dietary educational tools, is essential to enable meaningful improvements to be made to their health care. Educational psychologists report that adherence to any advice is improved when an individual's learning style (such as visual or auditory) and preferences for learning materials is provided for. Thus, although written or verbal explanations are the most common approaches, pictures and diagrams are more effective with visual learners. Similarly, adolescents report that they want more health-focused communications, presenting data as charts and graphs. In paediatric practice, the understanding of both the child and their parents must be considered and the parent-child interplay can influence the ability to learn. Sharing experiences and strategies between groups of parents and children can motivate long-term dietary changes. Healthcare professionals need to identify age-appropriate, relevant and engaging educational strategies informed by patient preferences, as these are most likely to empower, upskill and ensure optimal long-term adherence.

Rationale:

An international panel of paediatric renal dietitians and nephrologists from the Paediatric Renal Nutritional Taskforce (PRNT) have collaborated to develop a questionnaire (PUKA) to assess the baseline phosphate knowledge and understanding of CYP with CKD and their caregivers. A literature review was conducted to analyse existing instruments to evaluate phosphate knowledge. This showed that there was a lack of existing tools with proven validity and reliability that were suitable for use in paediatrics. However, this proved a useful guide for constructing a questionnaire and the questions chosen, format and design of the questionnaire was informed by those used in other studies, but expanded to gather background information on teaching preferences and problems experienced in relation to dietary changes or adherence to phosphate binder medication. This has been piloted on 10 CYP and their families to ensure face validity. The PUKA questionnaire will be completed by a purposive sample of CYP with CKD and caregivers in the 4 UK and 5 European nephrology units. The questionnaires will analysed to generate a phosphate knowledge score. Questions relating to personal opinions (such as preferred phosphate education approaches, perceived problems associated with implementing the reduced phosphate diet or taking phosphate binder medication) will be categorised and calculated as frequencies to represent the distribution of views. Correlation analysis will be used to measure the degree of association between any two variables (for example age, dialysis status, baseline biochemistry and knowledge score).

Current national and international PEM will be collated, evaluated and a representative sample selected. Focus groups of 5-6 children with CKD or caregivers will be run across these sites to gain feedback on these selected PEM and to further explore their perceived barriers and facilitators to adherence. The PUKA questionnaire and focus group data will be used to inform the development of PEM that address knowledge gaps and utilise the preferred education techniques. This novel approach will address adherence issues, empowering families to take ownership of phosphate management by personalising their child's care and offering patient choice, thereby optimising phosphate control and long-term bone and cardiovascular outcomes.

Benefits of research:

The investigators hope to find the real knowledge gaps and practical challenges experienced by CYP from diverse backgrounds, as represented across the partner sites to inform the co-design of PEM. Harnessing the expertise of an international team of dietitians and nephrologists is a unique strength of this proposal, including input from a clinical psychologist and 5 patient representatives. Patient-led resources will enable CYP to take control of their health, improve phosphate control and reduce long term adverse bone and cardiovascular outcomes. In addition, this project may also serve as a template to inform the development of future educational materials produced for children with kidney diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD4-5D between 8-18 years of age.
* One caregiver per patient.
* Consenting to study.

Exclusion Criteria:

* Children with neurodevelopmental or cognitive disorders.
* Children with an underlying phosphate-losing disease.
* Children on intensive dialysis regimens such as home haemodialysis or frequent daily in-centre HD.
* Children who are fully enterally tube fed.
* Children or caregivers with limited spoken or written language skills.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 50 caregiver-child dyads with CKD stage 4-5 and on dialysis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Characterise the facilitators and barriers to adherence to reduced dietary phosphate advice and phosphate binder medication administration in children and young people with CKD and their caregivers. | 2 years
  Qualitative - questionnaire and focus groups
Identify the preferred format and content of phosphate educational material of children and young people with CKD | 2 years
  Questionnaire and focus groups

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital for Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Palmer SC, Hayen A, Macaskill P, Pellegrini F, Craig JC, Elder GJ, Strippoli GF. Serum levels of phosphorus, parathyroid hormone, and calcium and risks of death and cardiovascular disease in individuals with chronic kidney disease: a systematic review and meta-analysis. JAMA. 2011 Mar 16;305(11):1119-27. doi: 10.1001/jama.2011.308. PMID 21406649
- [Background] Shroff R, Long DA, Shanahan C. Mechanistic insights into vascular calcification in CKD. J Am Soc Nephrol. 2013 Feb;24(2):179-89. doi: 10.1681/ASN.2011121191. Epub 2012 Nov 8. PMID 23138485
- [Background] Bertram JF, Goldstein SL, Pape L, Schaefer F, Shroff RC, Warady BA. Kidney disease in children: latest advances and remaining challenges. Nat Rev Nephrol. 2016 Mar;12(3):182-91. doi: 10.1038/nrneph.2015.219. Epub 2016 Feb 1. PMID 26831913
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD-MBD Update Work Group. KDIGO 2017 Clinical Practice Guideline Update for the Diagnosis, Evaluation, Prevention, and Treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD). Kidney Int Suppl (2011). 2017 Jul;7(1):1-59. doi: 10.1016/j.kisu.2017.04.001. Epub 2017 Jun 21. No abstract available. PMID 30675420
- [Background] McAlister L, Pugh P, Greenbaum L, Haffner D, Rees L, Anderson C, Desloovere A, Nelms C, Oosterveld M, Paglialonga F, Polderman N, Qizalbash L, Renken-Terhaerdt J, Tuokkola J, Warady B, Walle JV, Shaw V, Shroff R. The dietary management of calcium and phosphate in children with CKD stages 2-5 and on dialysis-clinical practice recommendation from the Pediatric Renal Nutrition Taskforce. Pediatr Nephrol. 2020 Mar;35(3):501-518. doi: 10.1007/s00467-019-04370-z. Epub 2019 Oct 30. PMID 31667620
- [Background] Farfan-Ruiz AC, Czikk D, Leidecker J, Ramsay T, McCormick B, Wilson K, Zimmerman D. Multidisciplinary Team versus a "Phosphate-Counting" App for Serum Phosphate Control: A Randomized Controlled Trial. Kidney360. 2020 Dec 15;2(2):290-297. doi: 10.34067/KID.0007132020. eCollection 2021 Feb 25. PMID 35373021
- [Background] Karamanidou C, Clatworthy J, Weinman J, Horne R. A systematic review of the prevalence and determinants of nonadherence to phosphate binding medication in patients with end-stage renal disease. BMC Nephrol. 2008 Jan 31;9:2. doi: 10.1186/1471-2369-9-2. PMID 18237373
- [Background] Hyperphosphataemia in chronic kidney disease: Evidence Update December 2014: A summary of selected new evidence relevant to NICE clinical guideline 157 'Management of hyperphosphataemia in patients with stage 4 or 5 chronic kidney disease' (2013) [Internet]. London: National Institute for Health and Care Excellence (NICE); 2014. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK552051/ PMID 31886981
- [Background] Abercrombie EL, Greenbaum LA, Baxter DH, Hopkins B. Effect of intensified diet education on serum phosphorus and knowledge of pediatric peritoneal dialysis patients. J Ren Nutr. 2010 May;20(3):193-8. doi: 10.1053/j.jrn.2009.10.011. Epub 2010 Mar 19. PMID 20303791
- [Background] Ahlenstiel T, Pape L, Ehrich JH, Kuhlmann MK. Self-adjustment of phosphate binder dose to meal phosphorus content improves management of hyperphosphataemia in children with chronic kidney disease. Nephrol Dial Transplant. 2010 Oct;25(10):3241-9. doi: 10.1093/ndt/gfq161. Epub 2010 Mar 22. PMID 20308040